CLINICAL TRIAL: NCT04160299
Title: Effectiveness of Alternative Therapy for Improving Cognition, Balance, and Physical Activity in Older Adults With Mild Cognitive Deficits for Home or Community-based Translation
Brief Title: Effectiveness of Alternative Therapy for Improving Cognition, Balance, and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tanvi Bhatt, Associate Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-1074; P30AG022849 (NIH)
Record Dates: First submitted 2019-09-09; First posted 2019-11-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment; Older Adults; Neurological Injury
MeSH Terms: conditions — Cognitive Dysfunction; Trauma, Nervous System | interventions — Dance Therapy

STUDY DESIGN:
Intervention Model Description: Older adults with Mild Cognitive Impairments, MCI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dance-based exergaming (Experimental): This will be an intervention-based study with single-group design, where participants will receive VR-based dance training for ten weeks. An anticipated 20 participants with a diagnosis of mild cognitive deficits will be recruited for initial screening
  Interventions: Behavioral: Dance-based exergaming

INTERVENTIONS:
Behavioral: Dance-based exergaming — Dance sessions
  Other Names: Dance therapy; Dance-based virtual reality

SUMMARY:
The composite effect of reduced balance, cognition, gait abnormalities/gait disturbances, and physical activity in older adults with mild cognitive impairments (MCI) leads to fear of falling and reduced participation in daily activities, which results in reduced cardiovascular fitness and deconditioning. Although many conventional balance and strength training programs have been implemented for older adults with MCI; these adults do not receive adequate practice dosage to make significant improvements, most likely due to lack of adherence to therapy and/or inadequate incorporation of all domains of the ICF model (body functions and structures, activities and participation) and lack of targeting cognitive-motor interference (deterioration of motor and/or cognitive function when both tasks are performed together). The use of alternative therapies such as dance and virtual reality (VR) has been found to be relatively enjoyable for older adults due to increased motivation, which led to the added improvement of physical and cognitive functioning. The overall aims of this pilot is to test the feasibility of VR-based dance therapy paradigm for older adults with MCI as well as its effect on enhancing balance, gait, and cognition, and physical fitness. Investigators also hope that the net effect of improvement in these domains of health outcomes will result in pre and post reduction of fall risk and improved quality of life of older adults with MCI.

The study investigates the effectiveness of a VR (Kinect)-based dance therapy in older adults with MCI by demonstrating its feasibility and compliance rate and also determine the efficacy of the VR-based dance therapy in improving health outcomes such as motor and cognitive functions, thereby reducing cognitive-motor interference. The study will also aim to determine the effectiveness of the VR-based dance paradigm in improving cardiovascular fitness and physical activity (PA) in older adults with MCI

DETAILED DESCRIPTION:
Aging results in neuromuscular deterioration, such as impaired balance control, gait instability, and worsening cognition, with increasing evidence pointing to the over-reliance on cognitive function to perform even simple motor tasks. Such deterioration has been shown to affect daily functional activities, quality of life, and cardiovascular fitness, along with an increase in the risk of falling. Recent literature has indicated that individuals with mild cognitive impairment (MCI) exhibit reduced gait speed during dual-tasking (DT) (performing a motor and cognitive task concurrently), thereby increasing the risk of falls. Physical activity has been recommended as a means to slow down neuromuscular deterioration and enhance gait, stability, and cognition in older adults with MCI. Further, increased levels of physical activity have also demonstrated positive effects on cardiovascular fitness (heart rate variability, HRV). However, older adults with MCI do not meet the recommended daily requirement (of at least 5000 steps/day) due to reduced motivation and lack of compliance to physical activity regimen. The lack of compliance may emanate from reduced levels of multisensory feedback, lack of involvement, and the decreased participatory nature of most conventional physical therapy interventions. As a result, there is the need to implement an alternative intervention for older adults with MCI. This alternative therapy should be motivational and enjoyable with increased participation or involvement, while providing increased sensorimotor feedback, and aiming to improve cognition, physical activity and balance for fall prevention in older adults. Dance therapy, as an alternative therapy, has shown to increase both physical and cognitive function as well as increase motivation among older adults. A preliminary study conducted with virtual reality (VR)-based dance, showed the integration of virtual reality and dance to be feasible in improving physical function and balance in people with stroke. It is postulated that people with MCI could benefit from an integrated VR-based dance therapy. However, there is no data on the feasibility and effect of VR-based dance therapy on compliance, cognitive, gait and physical activity measures among adults with MCI. Investigators, therefore, seek to examine the feasibility of alternative VR-based dance therapy through the use of commercially available and cost-effective Kinect systems in the laboratory setting. The reduced feasibility and lack of compliance associated with various forms of conventional therapy in MCI adults, due to reduced motivation, have been well documented. Dance, as an alternative therapy has been found to be more enjoyable while providing increased motivation for older adults, due to its effects on motivational brain centers of the nervous system. Dance stimulates interacting active brain centers that help in motor control, ambulation, and cognitive functions. Few studies have indicated that dance- based training activates Action Observation Network system (AON) and other brain centers, which is known to improve balance control through increased plasticity of neural systems (mirror neurons) for optimal observation and actual performance of dance. Impairment in cognitive function is depicted as slow gait during dual-task conditions. Slow gait dual tasking is relevant predictor of falls in older adults with MCI.

3.0 Objectives/Aims

Aim 1: To demonstrate feasibility and compliance rate of a VR-based dance training paradigm for community-based older adults with mild-cognitive impairment (CB-MCI). Hypothesis 1: At post-training, results will demonstrate feasibility of a VR-based dance therapy, which will be evaluated through both structured patient interviews and structured questionnaires [ITC-Sense of Presence Inventory questionnaire]. Participants will also demonstrate appropriate compliance (attend >24/30 session) and motivation (>Intrinsic Motivation Inventory scores) post-intervention.

Aim 2: To determine the effectiveness of VR-based dance training paradigm in improving motor and cognitive functions, by reducing cognitive-motor interference.

Hypothesis 2: When post-training tests are compared to those of pre-training, there will be a significant improvement in balance (on limits of stability test) and gait (in spatiotemporal parameters), motor and cognition (assessed by a neuropsychological test battery), which will result in overall reduced cognitive-motor interference (dual-task cost during balance and gait tasks).

Aim 3: To determine the effect of a VR-based dance training paradigm on improving cardiovascular (heart rate variability HRV) and physical fitness (physical activity, PA) of community-based older adults with MCI.

Hypothesis 3: Post-training measures will depict a significant improvement in cardiovascular and physical activity fitness.

Ancillary hypothesis (Aims 1-3): To determine if improved cognitive-motor function and physical fitness gained from a VR-based dance intervention will translate into improved fall efficacy and quality of life post withdrawal of intervention. Hypothesis: At 14 weeks (4 weeks post-intervention or withdrawal), participants will have retention of the post-training gains in cognitive-motor function and cardiovascular fitness, which will translate into improved falls efficacy (improvement on Activities-specific Balance Confidence scale), quality of life (Older People's Quality of Life Questionnaire (OPQOL-35) and participation (improved Community Integration Scale) compared to their pre-training.

Participants with MCI (≥ 65 years) will receive VR-based dance training for 10-weeks (30 sessions total) using the commercially available Kinect dance video game "Just Dance 3". Ten weeks of VR-based dance therapy falls within the normal duration for most dance and other alternative therapy studies provided for older adults. If successful, such intervention could then be implemented in the home or community setting and can then be delivered by caregivers either in an independent or assisted living facility after the caregivers receive training from the rehabilitation therapists.

ELIGIBILITY:
Inclusion Criteria:

* Age group: ≥65 years
* Montreal cognitive Assessment (MOCA) score <26/30
* Bone density with a t-score ≥ -2
* Absence of any acute or chronic neurological, cardiopulmonary, musculoskeletal, or systemic diagnosis.
* No recent major surgery (< 6 months)
* No recent hospitalization (< 3 months)
* Not on any sedative drugs
* Can understand and communicate in English

Exclusion Criteria:

* HR > 85% of age-predicted maximal heart rate (HRmax = 220 - age)
* Systolic blood pressure (SBP) > 165 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg during resting
* Oxygen saturation (measured by pulse oximeter) during resting < 95%
* Inability to stand for at least 5 minutes without an assistive device (length of dance game)
* History of bone fracture or significant other systemic disease or surgery in the last six months

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of a 10-week Virtual reality-based dance training: questionnaire | Week 10
  Feasibility of this pilot study will be determined by a feasibility questionnaire based on the ITC-Sense of Presence Inventory questionnaire. The ITC-Sense of Presence Inventory Questionnaire consists of questions and statements about the feasibility of the study and will be scored from 1(strongly disagree) to 5 (strongly agree). The questionnaire comprises of inputs regarding the participants' experiences in the virtual environment including perception and sense of presence in the virtual environment and about their experiences in the VR-based dance training environment, the presence of potential side effects and their input on the design and effects of the intervention.
Compliance rate of participants to a 10-week virtual reality-based dance training | End of all dance training sessions at Week 10
  Percentage of the number of sessions completed out of a total of 30 by each participant.
Change in cognitive functions during single and dual tasks | Baseline at Week 0, Mid-intervention at week 5, post-intervention week 11 and Follow-up at week 14
  Accuracy of performance to cognitive task which assesses attention, executive function and reaction time by the use of computerized Neuropsychological Battery test.
  Accuracy and reaction time will also be tested by serial subtraction, letter number sequence, Trial Making Test and category naming task. Performance and cost will be evaluated during dual tasking with Serial subtraction, letter number sequence and category fluency cognitive task while walking on gait rite, performing slip and trip test and also during volitional Limits of Stability, LOS and Sensory Organization Test, SOT with NeuroCoM Balance Master.
  Accuracy (number of correct responses out of the total responses). Higher accuracy indicates better performance.
Change in incidence of falls | Baseline at week 0 and Follow-up at week 14
  Change in the number of falls over 14 weeks will be assessed by the Fall Incidence Questionnaire. This fall questionnaire ascertains the number of falls experienced by participants over 14 weeks of the study. Reduction in the number of falls is a good indication of effectiveness of the intervention.
Change in end point excursion | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  It is the magnitude of a self-initiated movement (i.e., how far he/she wills to reach a target) without taking a step or losing balance measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Change in Movement velocity | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  It is the average speed of center of gravity movement during intentional movement measured in degrees per second under single and dual-task conditions. Higher values indicate better performance.
Change in maximum excursion | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  It is the actual magnitude of a self-initiated movement (i.e., how far did he/she actually reach a target) without taking a step or losing balance measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Change in directional control | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  It is the quality of a self-initiated movement (i.e., amount of movement actually exhibited towards the target to the amount of extraneous movement away from the target) measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Change in postural stability during reactive balance control (single and dual-task) | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Reactive stability balance, in terms of center of mass position and velocity during slips and trips will be assessed with ActiveStep Treadmill equipment and inertial sensors. Postural stability can be defined as simultaneous control of center of mass (COM) position and velocity during slip-like or trip like perturbation relative to the rear edge of base of support (rear heel). The position is normalized with the individual's foot length, and velocity by square root of gravitational acceleration and individual's body height. Larger values indicate greater stability.
Change in step length | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Step length (meters), which is a determinant of fall will be assessed with Gaitrite and inertial sensors.
Change in gait speed | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Gait speed (meters per second), which is determinant of fall will be assessed with Gaitrite and inertial sensors.
Change in cadence | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Cadence (steps per minute), which is determinant of fall will be assessed with Gaitrite and inertial sensors.

SECONDARY OUTCOMES:
Change in Blood pressure (mmHg) | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Blood pressure will be monitored during the course of the dance training in order to determine if there is any change in systolic or diastolic blood pressure. Change in heart rate will also be monitored in order to determine consistency in its variability, Heart rate variability, HRV.
Change in heart rate (beats per minute, bpm) | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Change in heart rate will also be monitored in order to determine consistency in its variability, Heart rate variability, HRV.
Change in physical activity level (step count) | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Change in step count before, during and after dance training will assessed by use of physical activity application (Health app on iPhone or Fit on Android) installed on smart phone. We shall also corroborate this data by assessing step count and other daily activities with Physical Activity Scale for the Elderly (PASE). Physical Activity Scale for the Elderly uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity.
Change in distance covered in Six-minute walk test (6MWT) | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Change in distance (in meters) covered during the performance of a 6MWT. The 6MWT assesses aerobic capacity and endurance of participants, with a normalized distance for older adult set between 392 and 572 meters.
Change in time taken to complete Timed-Up and Go (TUG) | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Change in time (in seconds) taken to complete TUG will provide us information about participants' mobility and balance statuses, as well fall risk. A score of between 7 and 12 seconds will be considered as the normal time for older adults to complete a TUG.
Berg Balance scale | Baseline at week 0, mid-intervention at week 5, post-intervention at week 11 and follow-up test at week 14
  Assess static and dynamic balance. This scale consists of the participant transferring from one chair to another, reaching forward, stepping up and down from a stepping stool, standing with eyes closed and open, one leg standing. It is a 14-item scale with each item score ranging from 0-4. Performance on the scale will be calculated on a total of 56. Less than 45 will indicate greater risk of falling.
Change in fall incidence in the home and community setting | Follow-up test at week 14
  At 4-week follow-up session, change in fall incidence will be assessed by Fall Incidence Questionnaire. This questionnaire determines the number of falls encountered by participants over the course of 14.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi Bhatt, PhD, Principal Investigator — University of Illinois at Chicago; Ernest K Ofori, MS, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data with concerned researchers stated in the IRB
Supporting Information: Study Protocol, SAP, ICF
Time Frame: November 2018 - December 2020